CLINICAL TRIAL: NCT03616145
Title: Effects of Osteopathic Manipulative Treatment (OMT) on Gait Biomechanics in Parkinson's Disease (OMT/PD)
Brief Title: Effects of Osteopathic Manipulative Treatment (OMT) on Gait Biomechanics in Parkinson's Disease
Acronym: (OMT/PD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Hollis King, Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13517128719
Record Dates: First submitted 2018-07-04; First posted 2018-08-06 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Parkinson Disease
Keywords: Osteopathic Manipulative Treatment
MeSH Terms: conditions — Parkinson Disease | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: The overall design proposed in this study is a randomized, placebo controlled, single-blind controlled trial. Data will be collected in this developmental study to assess potential differences in gait, balance, and quality of life of patients in the intervention arm (6-week OMT intervention coupled with standard of care (SOC) versus the light touch comparator arm (6-week light touch coupled with SOC) versus the non-intervention control arm (SOC alone).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding. The PI, statistician, recruitment personnel, research assistants conducting the assessment sessions, and data entry/verification clerks will be blind to participant's group assignment until data is unlocked at the end of the study. Only the Project Manager who will develop and oversee the randomization procedure, prepare progress reports, and inform participants of their treatment condition will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Osteopathic Manipulative Treatment (OMT) (Experimental): Participants assigned to the OMT arm will receive 6 weekly sessions. The provider will perform the following 14 osteopathic procedures 1) lateral (and anteroposterior) translation of vertebrae in the thoracic/lumbar spine; 2) active myofascial stretch to the thoracic spine; 3) occipito-atlanto release; 4) translation of cervical spine; 5) muscle energy techniques of the cervical spine; 6) Spencer technique applied to the shoulder bilaterally; 7) supination/pronation of the forearm; 8) circumduction of the wrist; 9) sacroiliac joint gapping; 10) muscle energy technique applied to adductor muscles of lower extremity; 11) psoas muscle energy technique; 12) hamstring muscle energy technique; 13) articulatory technique applied to the ankle; 14) and muscle energy technique applied to the ankle in dorsi and plantar flexion. Further, each subject will receive cranial assessment and treatment emphasizing the venous sinus techniques and compression of the fourth ventricle (CV-4).
  Interventions: Procedure: Osteopathic Manipulative Treatment (OMT)
- Light Touch (Sham Comparator): Participants assigned to the light touch comparator arm will receive 30 minutes of light touch procedures designed to be credible but minimally effective. The procedures for the light touch arm are adapted from the methodology established in the North Texas Chronic Low Back Pain Trial, and have been used successfully by the PI as a comparator arm numerous times in the past (e.g., in the OSTEPAThic Trial). Subjects assigned to receive light touch will be treated in positions similar to subjects receiving OMT. Light touch will target each of the 15+ anatomic regions for approximately 1 ½ to 2 minutes each to appropriately control for time, attention, and physical contact. Light touch hand placement will be over the same areas of the body contacted in the OMT protocol, but involve virtually no motion of a meaningful nature, such a range of motion testing which could have therapeutic effect.
  Interventions: Other: Light Touch
- Standard of Care Only (No Intervention): Subjects will continue their usual care and will visit the UCSD for the 4 assessment sessions only, during their course of study participation.

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment (OMT) — Experimental Condition
  Arms: Osteopathic Manipulative Treatment (OMT)
Other: Light Touch — Comparator Arm
  Arms: Light Touch

SUMMARY:
Parkinson's disease (PD) is a neurological disorder that puts individuals at high risk for injuries and long-term disabilities as a result of a fall or other trauma. Injuries sustained from falls account for many deaths as well as thousands of hospital admissions and nursing home stays every month. Quality of life and even longevity itself is reduced due to the resulting surgeries, immobility, complications and even cognitive impairments that can follow. The proposed study will explore beneficial impact of a treatment modality (OMM/OMT) that may significantly reduce the morbidity of this condition by comparing 6 weeks of OMT versus 6 weeks light touch intervention versus 6 weeks care as usual to improve gait in individuals with PD. Gait will be measured at mid-treatment, post-treatment and 4-week follow-up.

DETAILED DESCRIPTION:
The overall design proposed in this study is a randomized, placebo controlled, single-blind controlled trial. Data will be collected in this developmental study to assess potential differences in gait, balance, and quality of life of patients in the intervention arm (6-week OMT intervention coupled with standard of care (SOC) versus the light touch comparator arm (6-week light touch coupled with SOC) versus the non-intervention control arm (SOC alone). As noted in the previous section, power analyses assuming a clinically significant improvement in gait and balance indicate that 90 completers per condition will be enough to detect this medium effect size. To achieve this aim, the investigators will over-recruit to allow for ~20% dropout rate by recruiting a total of 108 participants (36 per condition). The benefit of OMT as compared to standard care for PD is what is being examined in this study and if shown beneficial may be a less invasive with fewer side effects that standard care which may utilize surgery.

Randomization will occur after baseline testing session. Individuals will be randomly assigned to one of three treatment arms using a computer-generated randomization algorithm that will determine group assignment in variable blocks of 3 & 6 and stratified by gender. Study staff completing the assessment sessions will remain naive to treatment condition. All study staff will be CITI-certified prior to study commencement.

The 6 OMT and the light touch comparator arm sessions will be administered at the UCSD EPARC offices, or at Osteopathic Center San Diego.

OMT Intervention Arm. Along with SOC, participants assigned to the OMT arm will receive 30 minutes of OMT per week for 6 weeks. Following the precedent of OMT procedures used by Wells et al., (1999), the provider will perform the following 14 osteopathic procedures 1) lateral (and anteroposterior) translation of vertebrae in the thoracic/lumbar spine; 2) active myofascial stretch to the thoracic spine; 3) occipito-atlanto release; 4) translation of cervical spine; 5) muscle energy techniques of the cervical spine; 6) Spencer technique applied to the shoulder bilaterally; 7) supination/pronation of the forearm; 8) circumduction of the wrist; 9) sacroiliac joint gapping; 10) muscle energy technique applied to adductor muscles of lower extremity; 11) psoas muscle energy technique; 12) hamstring muscle energy technique; 13) articulatory technique applied to the ankle; 14) and muscle energy technique applied to the ankle in dorsi and plantar flexion. All of these OMT procedures are used in standard OMT practice and are gentle non-thrusting maneuvers in general. Further, each subject will receive cranial assessment and treatment emphasizing the venous sinus techniques and compression of the fourth ventricle (CV-4). The addition of the CV-4 beyond the 14 areas assessed and treated in the Wells et al study reflects research that showed CV-4 impact on sleep latency and muscle sympathetic activity impact on brain oxygen levels as well as alpha rhythm. The utilization of the venous sinus technique is based on its impact in increasing blood flow to the circle of Willis and Dr. King's pilot work. The myofascial and other appropriate OMT procedures are directed at the whole neuromusculoskeleton system and benefit postural balance and range of motion in general. Given the rare risk of spinal cord injury or vertebral artery dissection with high velocity, low amplitude techniques, these will not be utilized on this protocol. Participants undergoing OMT intervention will continue with their current standard of care.

Comparator Arm (Light Touch) : Participants assigned to the light touch comparator arm will receive 30 minutes of light touch procedures designed to be credible but minimally effective. The procedures for the light touch arm are adapted from the methodology established in the North Texas Chronic Low Back Pain Trial, and have been used successfully by the PI as a comparator arm numerous times in the past (e.g., in the OSTEPAThic Trial). Subjects assigned to receive light touch will be treated in positions similar to subjects receiving OMT. Light touch will target each of the 15+ anatomic regions for approximately 1 ½ to 2 minutes each to appropriately control for time, attention, and physical contact. Light touch hand placement will be over the same areas of the body contacted in the OMT protocol, but involve virtually no motion of a meaningful nature, such a range of motion testing which could have therapeutic effect. The subject will feel hand contact, a light touch, but no treatment intention expressed by the operator verbally or by hand motion. While the operator's hands will be placed of areas contacted in the OMT protocol, the precise placement will be off, away from, the real OMT procedures. The intent of the light touch is to apply manual forces of diminished magnitude purposely aimed to avoid treatable areas of somatic dysfunction relative to gait and balance dysfunction in PD and, consequently, to minimize the likelihood of any therapeutic effect.

Standard of Care (SOC) Only. Subjects will continue their usual care and will visit the UCSD for the 4 assessment sessions only, during their course of study participation.

After the 4-week follow-up assessment visit, all participants assigned to light touch or SOC arms will be offered the opportunity to receive 6 weeks of OMT, if they so desire.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Ambulatory without use of assistive device.
3. Fluency in written and spoken English.
4. Montreal Cognitive Assessment (MoCA) score > or = 17.
5. Stages 1 - 4 Parkinson's Disease diagnosis as measured by the Unified Parkinson's disease rating scale.

Exclusion Criteria:

1. Currently enrolled in another clinical trial.
2. Current taking PD medications co-morbid conditions such as pseudobulbar palsy or amyotrophic lateral sclerosis which may have musculoskeletal effects.
3. Individuals with current fractures, tumors, wounds.
4. Any lifetime Deep Brain Stimulation implant surgery.
5. Recent surgeries, eg., within past 90 days.
6. Patients who have experienced hospitalization due to a fall within the past 12 months.
7. Gait abnormalities other than Parkinson's disease.
8. Received OMT or another forms of manipulative therapy within the past two months.
9. Stage 5 Parkinson's Disease diagnosis per as measured by the Unified Parkinson's disease rating scale.
10. Other co-morbid conditions that in the opinion of the PI would interfere with participation in this study.
11. Diagnosis of psychosis or dementia (MoCA, DRS or other indication in eMR).
12. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 94 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2024-01-21 (Estimated)

PRIMARY OUTCOMES:
Change in Gait | 0 weeks, 6 weeks, and 10 weeks
  Gait analysis will be conducted using the Timed Up and Go while wearing the LEGsys+ system. The Legsys body worn sensor system utilizes state-of-the-art camera-based motion capture allowing measurement of advanced gait parameters including stride duration and length, step length, speed, cadence, sagittal plane knee and hip angles, and superior-inferior and medial-lateral pelvis movement, as well as a fall risk assessment.
Change in Balance | 0 weeks, 6 weeks, and 10 weeks
  Balance will be measured via the NeuroCom SMART EquiTest system, which enables enables the isolation and assessment of the sensory and muscular components of balance.

SECONDARY OUTCOMES:
Change in Cognition | 0 weeks, 6 weeks, and 10 weeks
  The Montreal Cognitive Assessment (MoCA) will be administered as a measure of general cognition and will be used as a covariate in the statistical analyses (please see Data Analysis section below). The MoCA is a suitably accurate, brief (10-minute) test of cognitive impairment in PD and has established cut-offs for both MCI and PDD.
Change in PD-Related Health Status | 0 weeks, 6 weeks, and 10 weeks
  Parkinson's Disease Questionnaire-39 (PDQ-39) is a self-report measure of health status (HS), which is considered different than QoL in that it does not ask for perceptions, judgments or reactions. It consists of 39 questions rated by the subject on a five-item likert scale (Never, Occasionally, Sometimes, Often, or Always) and takes approximately 10 minutes to complete. From these questions, eight subscale (Mobility, Activities of Daily Living, Emotional Well-Being, Stigma, Social Support, Cognition, Communications, and Bodily Discomfort) scores are derived by summing the item scores for each subscale, dividing the sum by the highest possible score for that subscale and then multiplying this number by 100. Higher scores correspond to worse HS.
Change in Depressed Mood | 0 weeks, 6 weeks, and 10 weeks
  Geriatric Depression Scale (GDS) is a self report questionnaire comprised of 30 yes or no questions used to identify depression in the elderly. Total scores range from 0 to 30 where higher scores reflect more severe depression 11 .
Change in Motor Skills | 0 weeks, 6 weeks, and 10 weeks
  The Movement Disorder Society-The Unified Parkinson's disease Rating Scale (MDS- UPDRS Part Three). For this assessment participants go through a series of tasks designed to assess various motor characteristics such as speech, facial expression, rigidity, finger tapping, hand movements, toe tapping, freezing of gait, etc. All scores for each component range from 0 to 4 and summed for a grand total 4

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No